CLINICAL TRIAL: NCT03687060
Title: Behavioral Economics and Implementation Research to Reduce Cardiovascular Risk in HIV-Infected Adults
Brief Title: INcreasing Statin Prescribing in HIV Behavioral Economics REsearch
Acronym: INSPIRE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of California, Los Angeles (Other)
Collaborators: RAND (Other); Olive View-UCLA Education & Research Institute (Other)
Responsible Party: Principal Investigator, Allison L. Diamant, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 1U01HL142104-01 (NIH)
Record Dates: First submitted 2018-09-20; First posted 2018-09-27 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: HIV; Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: Stepped-wedge cluster randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Organization Level (Other)
  Interventions: Behavioral: Knowledge assessment
- Provider Level (Other)
  Interventions: Behavioral: Knowledge assessment; Behavioral: Education Intervention; Behavioral: Provider Feedback
- Patient Level (Other)
  Interventions: Behavioral: Knowledge assessment

INTERVENTIONS:
Behavioral: Knowledge assessment — Investigators will conduct semi-structured interviews with medical directors, clinical leadership and all participating physicians to gain insight on knowledge about and barriers to prescribing statins for people living with HIV. People living with HIV will participate in focus groups.
Behavioral: Education Intervention — Education intervention will be adapted from the the findings of these interviews and focus groups.
  Clinics will be randomized to receive the "education intervention and feedback" implementation strategies at different times.
  Medical directors and providers will receive a brief educational intervention about cardiovascular disease risk in people living with HIV. Providers will additionally receive a web-based survey before and after the education intervention.
  Patients will receive pamphlets tailored to the effects of cardiovascular disease treatment for people living with HIV.
  Arms: Provider Level
Behavioral: Provider Feedback — Six months after the education intervention, providers will receive monthly emails with feedback regarding their rates of prescribing statins, with language targeted at increasing motivation to prescribe by leveraging social norms and self-image.
  Arms: Provider Level

SUMMARY:
Cardiovascular disease is a major cause of morbidity and mortality among people living with HIV. Recent studies have demonstrated that patients with HIV experience a 50-100% increased risk of myocardial infarction and stroke compared to HIV-uninfected persons. They also face higher risks of stroke, sudden death, and heart failure. However, evidence-based statin therapy-which is safe in this population and highly effective at reducing cardiovascular risk-is under-prescribed. The investigators propose a multi-level intervention to increase evidence-based statin prescribing by addressing barriers at these levels. The implementation intervention includes two strategies: (1) tailored education at the leadership, provider, and patient levels, and (2) behavioral economics-informed feedback for providers.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 40 years
* have been diagnosed with HIV
* LDL ≥ 190, diabetes and LDL ≥ 70
* or 10-year ASCVD risk ≥ 7.5%
* or history of heart attack, stroke, or peripheral vascular disease
* care for patients with HIV at least 1/2 day each week (physicians)
* work at participating clinics (physicians)

Exclusion Criteria:

* unable to provide written, informed consent
* not at participating clinic

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Change in proportion of PLWH with cardiovascular risk factors seen by a physician receiving statin therapy | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Allison Diamant, MD, MSHS, Principal Investigator — University of California, Los Angeles; William Cunningham, MD, MPH, Principal Investigator — University of California, Los Angeles
Locations (8):
- United States (8):
  - JWCH Institute, Commerce, California
  - Antelope Valley Health Center, Lancaster, California
  - Watts Health Center, Los Angeles, California
  - Oasis Clinic, Los Angeles, California
  - To Help Everyone Health and Wellness Centers, Los Angeles, California
  - Venice Family Clinic, Santa Monica, California
  - Olive View-UCLA Medical Center, Sylmar, California
  - Tarzana Treatment Centers, Inc., Tarzana, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Feinstein MJ, Bahiru E, Achenbach C, Longenecker CT, Hsue P, So-Armah K, Freiberg MS, Lloyd-Jones DM. Patterns of Cardiovascular Mortality for HIV-Infected Adults in the United States: 1999 to 2013. Am J Cardiol. 2016 Jan 15;117(2):214-20. doi: 10.1016/j.amjcard.2015.10.030. Epub 2015 Nov 6. PMID 26639041
- [Background] Aberg JA, Sponseller CA, Ward DJ, Kryzhanovski VA, Campbell SE, Thompson MA. Pitavastatin versus pravastatin in adults with HIV-1 infection and dyslipidaemia (INTREPID): 12 week and 52 week results of a phase 4, multicentre, randomised, double-blind, superiority trial. Lancet HIV. 2017 Jul;4(7):e284-e294. doi: 10.1016/S2352-3018(17)30075-9. Epub 2017 Apr 13. PMID 28416195
- [Background] Masia M, Bernal E, Robledano C, Padilla S, Lopez N, Martinez E, Gutierrez F. Long-term effects of an intensive intervention in HIV-infected patients with moderate-high atherosclerotic cardiovascular risk. J Antimicrob Chemother. 2014 Nov;69(11):3051-6. doi: 10.1093/jac/dku269. Epub 2014 Jul 18. PMID 25038306
- [Background] Freiberg MS, Chang CC, Kuller LH, Skanderson M, Lowy E, Kraemer KL, Butt AA, Bidwell Goetz M, Leaf D, Oursler KA, Rimland D, Rodriguez Barradas M, Brown S, Gibert C, McGinnis K, Crothers K, Sico J, Crane H, Warner A, Gottlieb S, Gottdiener J, Tracy RP, Budoff M, Watson C, Armah KA, Doebler D, Bryant K, Justice AC. HIV infection and the risk of acute myocardial infarction. JAMA Intern Med. 2013 Apr 22;173(8):614-22. doi: 10.1001/jamainternmed.2013.3728. PMID 23459863
- [Background] Stein JH. Management of Lipid Levels and Cardiovascular Disease in HIV-Infected Individuals: Just Give Them a Statin? Top Antivir Med. 2016 Dec-2017 Jan;23(5):169-73. PMID 27398770
- [Background] Thompson-Paul AM, Lichtenstein KA, Armon C, Palella FJ Jr, Skarbinski J, Chmiel JS, Hart R, Wei SC, Loustalot F, Brooks JT, Buchacz K. Cardiovascular Disease Risk Prediction in the HIV Outpatient Study. Clin Infect Dis. 2016 Dec 1;63(11):1508-1516. doi: 10.1093/cid/ciw615. Epub 2016 Sep 9. PMID 27613562
- [Background] Ladapo JA, Richards AK, DeWitt CM, Harawa NT, Shoptaw S, Cunningham WE, Mafi JN. Disparities in the Quality of Cardiovascular Care Between HIV-Infected Versus HIV-Uninfected Adults in the United States: A Cross-Sectional Study. J Am Heart Assoc. 2017 Nov 14;6(11):e007107. doi: 10.1161/JAHA.117.007107. PMID 29138182
- [Background] Jin J, Sklar GE, Min Sen Oh V, Chuen Li S. Factors affecting therapeutic compliance: A review from the patient's perspective. Ther Clin Risk Manag. 2008 Feb;4(1):269-86. doi: 10.2147/tcrm.s1458. PMID 18728716
- [Background] Lubloy A. Factors affecting the uptake of new medicines: a systematic literature review. BMC Health Serv Res. 2014 Oct 20;14:469. doi: 10.1186/1472-6963-14-469. PMID 25331607
- [Background] Doroodchi H, Abdolrasulnia M, Foster JA, Foster E, Turakhia MP, Skelding KA, Sagar K, Casebeer LL. Knowledge and attitudes of primary care physicians in the management of patients at risk for cardiovascular events. BMC Fam Pract. 2008 Jul 8;9:42. doi: 10.1186/1471-2296-9-42. PMID 18611255
- [Background] Trinkley KE, Malone DC, Nelson JA, Saseen JJ. Prescribing attitudes, behaviors and opinions regarding metformin for patients with diabetes: a focus group study. Ther Adv Chronic Dis. 2016 Sep;7(5):220-8. doi: 10.1177/2040622316657328. Epub 2016 Aug 11. PMID 27583122
- [Background] Cohen JD, Brinton EA, Ito MK, Jacobson TA. Understanding Statin Use in America and Gaps in Patient Education (USAGE): an internet-based survey of 10,138 current and former statin users. J Clin Lipidol. 2012 May-Jun;6(3):208-15. doi: 10.1016/j.jacl.2012.03.003. PMID 22658145
- [Background] Fung V, Sinclair F, Wang H, Dailey D, Hsu J, Shaber R. Patients' perspectives on nonadherence to statin therapy: a focus-group study. Perm J. 2010 Spring;14(1):4-10. doi: 10.7812/tpp/09-090. PMID 20740125
- [Background] Wei MY, Ito MK, Cohen JD, Brinton EA, Jacobson TA. Predictors of statin adherence, switching, and discontinuation in the USAGE survey: understanding the use of statins in America and gaps in patient education. J Clin Lipidol. 2013 Sep-Oct;7(5):472-83. doi: 10.1016/j.jacl.2013.03.001. Epub 2013 Mar 13. PMID 24079289
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] Aarons GA. Mental health provider attitudes toward adoption of evidence-based practice: the Evidence-Based Practice Attitude Scale (EBPAS). Ment Health Serv Res. 2004 Jun;6(2):61-74. doi: 10.1023/b:mhsr.0000024351.12294.65. PMID 15224451
- [Background] Lehman WE, Greener JM, Simpson DD. Assessing organizational readiness for change. J Subst Abuse Treat. 2002 Jun;22(4):197-209. doi: 10.1016/s0740-5472(02)00233-7. PMID 12072164
- [Background] Glisson C, Landsverk J, Schoenwald S, Kelleher K, Hoagwood KE, Mayberg S, Green P; Research Network on Youth Mental Health. Assessing the organizational social context (OSC) of mental health services: implications for research and practice. Adm Policy Ment Health. 2008 Mar;35(1-2):98-113. doi: 10.1007/s10488-007-0148-5. Epub 2007 Dec 18. PMID 18085434
- [Background] Weiner BJ, Amick H, Lee SY. Conceptualization and measurement of organizational readiness for change: a review of the literature in health services research and other fields. Med Care Res Rev. 2008 Aug;65(4):379-436. doi: 10.1177/1077558708317802. Epub 2008 May 29. PMID 18511812